CLINICAL TRIAL: NCT02361918
Title: Predicting Value of Serum Procalcitonin, C-reactive Protein, and Drain Fluid Culture, Fluid Il-6 and Tnf-α Levels in Anastomotic Leakage Following Rectal Resection
Brief Title: Predictive Value of Procalcitonin, CRP, Drain Fluid Culture, Il-6 and Tnf-α in Anastomotic Leakage
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Engin HATIPOGLU, M.D., Istanbul University
Other Study IDs: CTF-EH0001
Record Dates: First submitted 2014-10-26; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Anastomotic Leakage in Colon Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Anastomotic leakage: Patient had anastomotic leakage
  Interventions: Procedure: Colon surgery
- No anastomotic leakage: Patient had no anastomotic leakage
  Interventions: Procedure: Colon surgery

INTERVENTIONS:
Procedure: Colon surgery

SUMMARY:
Evaluating predictive value of serum procalcitonin, C-Reactive Protein, drain IL-6 and TNF-alpha for anastomotic leakage in post-operative period.

DETAILED DESCRIPTION:
To search for a biomarker, which might be able to predict rectal anastomotic leakage before its clinical presentation. Serum procalcitonin, C-reactive protein, and drain fluid culture, IL-6 and TNF-α levels were evaluated in 50 consecutive patients with rectal cancer who underwent low anterior resection with colorectal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent to colonic resection and had drain

Exclusion Criteria:

* other patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient had colonic resection
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Predictive values of serum CRP, procalcitonin, drain fluid IL-6 and TNF-alpha levels in anastomotic leakage. | 5 day